CLINICAL TRIAL: NCT05582616
Title: The Safety and Feasibility of Transcranial Direct Current Stimulation Combined With Conservative Treatment for Cervicogenic Headaches
Brief Title: The Safety and Feasibility of tDCS Combined With Conservative Treatment for Cervicogenic Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB22-0890
Record Dates: First submitted 2022-08-22; First posted 2022-10-17 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-01

CONDITIONS: Cervicogenic Headache
Keywords: Transcranial Direct Current Stimulation; Physiotherapy
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Double blind randomized placebo controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, researcher, and care providers will be blinded until after the analysis period, researchers will be assessing outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS with physiotherapy (Experimental): Patients will engage in a six-week treatment protocol with 3 sessions per week (18 treatments). This was chosen to minimize discomfort and ensure the number of sessions is consistent with previous migraine literature. The primary motor cortex (M1) will be the treatment target to reduce pain sensitivity and improve motor learning. M1 will be found through measurements of the head: the point halfway between the nasion and inion and halfway between the left and right tragus will be found, we will then move down 20% of the inter-tragi distance and place the anode there. The cathode will then be placed over the super orbital region. Each electrode will be held in place with a strap and will make as much contact with the skin as possible. tDCS will be delivered via two 35cm2 surface sponge electrodes at an intensity of 2mA in the active group.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS with physiotherapy (Sham Comparator): In the sham condition, the number of sessions, placement of electrodes, and types of electrodes used will be the same, however, only a 30 second ramp up period will be administered to emulate active tDCS therapy. Patients will be able to hear the sounds of the device and will feel slight tingling for the first 30 seconds but will receive no active stimulation. Previous sham studies have demonstrated efficacy of the blinding method.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — See treatment arm description
  Arms: Active tDCS with physiotherapy
Device: Sham Transcranial Direct Current Stimulation — See sham comparator arm description
  Arms: Sham tDCS with physiotherapy

SUMMARY:
Annually, up to 150,000 individuals are affected by cervicogenic headaches (CGH) in Canada with many of these cases being chronic. Current treatments for CGH are limited in efficacy and durability - indicating a dire need for novel interventions in this population. Transcranial direct current stimulation (tDCS) and physiotherapy have a high degree of safety and have been studied as interventions for many other chronic pain conditions and headache disorders. We propose to study the feasibility and safety of tDCS alongside physiotherapy for CGH further in a randomized sham controlled trial.

DETAILED DESCRIPTION:
Annually, up to 150,000 people in Canada and experience cervicogenic headaches (CGH) with many of these patients suffering from chronic CGH. CGH is a pain disorder where pain is perceived in the head but caused by dysfunction of the cervical spine and its anatomical structure. More specifically, the pathogenesis of CGH is due to the convergence of nociceptive afferents from the upper three cervical nerves and trigeminal nerves onto second-order neurons in the trigeminocervical nucleus. The pain signaling resulting from this is also modulated through sensorineural pathways involving the thalamus and the sensorimotor cortex. As such symptoms of CGH include restricted movement, local tenderness of the upper cervical spine joints, musculoskeletal impairments, headache, local pressure hyperalgesia and bilateral thermal hypoesthesia. To date, there is no "cure" for chronic CGH and current treatment entails trial and error with behavior management, environmental modifications and medications. Consequently, there is a significant need for new approaches to symptom management in order to help improve functional impairment and disease burden associated with treating CGH. Transcranial direct current stimulation (tDCS) and physiotherapy have a high degree of safety and have been studied as an intervention for many other chronic pain conditions and headache disorders, including arthritis and migraines, demonstrating considerable potential. The investigators propose to study the safety and feasibility of tDCS alongside physiotherapy as a treatment for CGH in a randomized sham controlled trial.

RESEARCH QUESTIONS AND OBJECTIVES

The overall objective is to study the feasibility and safety of tDCS applied to the primary motor cortex in patients with CGH and to explore whether active tDCS augments the effect of rehabilitation therapy.

Specifically the objectives are:

Primary Objective: To determine whether active tDCS is feasible and safe compared to sham when administered with rehabilitation therapy for patients with CGH when administered 3 times per week over the course of 6 weeks. Safety will be measured through serious adverse events (defined as events requiring medical attention). Feasibility will be measured by recruitment (greater than 30%), retention (greater than 80%), and adherence (greater than 70%). These outcomes will be measured throughout the treatment process up to immediately post-treatment.

Secondary Objective: To determine what secondary outcomes such as quality of life, headaches, pain sensitivity, neck mobility, anxiety, and depression improve with active tDCS treatment in individuals suffering with CGH. Quality of life will be measured via the European Quality of Life Five Dimension (EQ-5D), headache intensity, frequency, duration, and impacts on life will be measured via headache diaries and the Headache Intensity Test - 6 (HIT-6), headache effects on participant function will be measured via the Headache Disability Index (HDI), neck pain intensity will be measured through the numeric pain rating scale (NPRS), pain sensitivity will be measured via the Pain Sensitivity Questionnaire (PSQ), pain impacts on quality of life will be measured through the patient reported outcomes measurement information system - pain interference scale (PROMIS-PI), neck mobility will be measured through various motor control, strength, and endurance tests, feelings of depression will be measured via the PHQ-9 and anxiety via the GADS-7 before treatment after treatment and at 6- and 12- weeks post treatment.

Third objective: To explore whether the effects of active tDCS will augment the effects of rehabilitation therapy in treating individuals with CGH.

METHODS

This study will be a double-blind, sham-controlled, concealed allocation, randomized, clinical trial.

Clinical Assessments: Demographic information will be collected two weeks prior to starting the study including age, sex, education, headache history, concussion history, past medical history, medication use, and family medical history. Baseline questionnaires will be completed including 2-weeks of Headache Diaries Headache Impact Test - 6 (HIT-6), Rivermead PPCS questionnaire (RPQ), Headache Disability Index (HDI), European Quality of Life Five Dimension (EQ-5D), patient health questionnaire-9 (PHQ-9), generalized anxiety disorder scale-7 (GADS-7), Patient Reported Outcomes Measurement Information System Pain Interference Sub-scale (PROMIS-PI), the Pain Catastrophizing Scale (PCS), and the Numeric Pain Rating Scale (NPRS). Furthermore the following baseline neck mobility assessments will be used: the Craniocervical Flexion Test (CCFT), the Cervical Extensor Endurance Test (CEET), the Dynamometry Neck-Strength Assessment (DNSA), a range of cervical motion assessment (ROM), and a manual examination of the cervical joints (MECJ). Patients will keep a two-week baseline headache diary before treatment, 2 weeks during treatment, 2 weeks following tDCS, and for 2 weeks before the 6 and 12 week follow up assessments (total of 8 weeks). Patients will be reassessed at the completion of their tDCS treatment, and at 6- and 12-weeks post-treatment. The assessments administered at each follow up are: 2-week Headache Diaries, RPQ, HIT-6, HDI, EQ-5D, PHQ-9, GAD-7, NPRS, PCS, PROMIS-PI, CCFT, CEET, DNSA, ROM, and MECJ.

tDCS Protocol: Patients will engage in a six-week treatment protocol with 3 sessions per week (18 treatments). This was chosen to give participants at least a day between each session in order to minimize discomfort and because the number of sessions is consistent with previous migraine literature. The primary motor cortex (M1) will be the treatment target given previous literature highlighting reduced pain sensitivity and improved motor learning outcomes following tDCS stimulation of this region. M1 will be found through measurements of the head; more specifically the point halfway between the nasion and inion as well as halfway between the left and right tragus will be found, from here we will move down 20% of the distance between the left and right tragus while staying on the line between tragi. The anode will be placed over the M1 while the cathode will be placed over the super orbital region; each electrode will be held in place with a strap and will make as much contact with the skin as possible. tDCS will be delivered via two 35cm2 surface sponge electrodes at an intensity of 2mA in the active group and 0mA in the sham group. There will be a 30 second fade in and fade out period before and after stimulation with 20 minutes of active stimulation. In the sham condition, participants will only experience the 30 second fade in period and then the stimulator will be turned off. Previous sham studies have demonstrated the efficacy of this blinding method.

Physiotherapy Protocol: Participants will engage in a six-week physiotherapy program which will occur immediately following each tDCS session. The exercises to be used focus on head and back strength and motor control and were assembled by a licensed physiotherapist based on previous physiotherapy protocols for treating CGH. The exercises are performed at a level that is pain-free and are progressed when goals are reached (approximately every 2 weeks). Participants will also be expected to increase daily physical activity levels to 30 minutes per day for at least 5 days a week as a part of the physiotherapy program. This will be tracked using an exercise diary to be completed by participants each day.

Statistical Analysis: Summary statistics will be done and reported so that feasibility and safety can be assessed and future studies can use the results presented for power calculations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervicogenic headaches based on International Headache Society Guidelines lasting greater than 12 weeks
* The International Headache Society Guidelines are as follows: A) Presence of a headache fulfilling criterion C; B) Clinical and/or imaging evidence of a disorder or lesion within the cervical spine or soft tissues of the neck, known to be able to cause headache; C) Evidence of causation demonstrated by at least two of the following: (a) Headache has developed in temporal relation to the onset of the cervical disorder or appearance of the lesion; (b) Headache has significantly improved or resolved in parallel with improvement in or resolution of the cervical disorder or lesion; (c) Cervical range of motion is reduced and headache is made significantly worse by provocative maneuvers; (d) Headache is abolished following diagnostic blockade of a cervical structure or its nerve supply.
* Average pain score ≥ 4/10 and Neck Disability score ≥ 28/50

Exclusion Criteria:

* Known cervical spine pathology (such as tumours or fractures)
* Nerve root pain/sensory loss
* Muscular or joint inflammatory conditions
* Neurological or psychiatric conditions
* Undergone recent surgery (within prior year)
* Have contraindications to tDCS (metal or electronic implants in the brain/skull; metal or electronic implants in other sites on the body; surgical procedures involving the head or spinal cord; skin problems such as dermatitis, psoriasis or eczema; epilepsy or a previous convulsion/seizure; fainting spells or syncope; pregnancy or any chance of pregnancy; previous electrical or magnetic stimulation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Feasibility of tDCS through recruitment rate, retention rate in the study, and adherence rates to both tDCS and exercise therapy. | To be assessed throughout the 6 weeks of treatment and at post-treatment follow-up.
  The feasibility of tDCS will be measured through the rate of participants contacted vs those actually enrolled (expected to be greater than 30%), through rate of those enrolled vs those completing 6-weeks of treatment (expected to be greater than 80% retained), and through rates of those who completed all 18 tDCS sessions in 6-weeks as well as the percentage of exercise therapy sessions completed within the 6-week study period (expected to be greater than 70% for both).
Safety of tDCS through adverse events and transient changes in adverse effects within each tDCS session. | To be assessed throughout the 6 weeks of treatment up to the post-treatment follow-up.
  The safety of tDCS will primarily be measured through tracking rates of serious adverse effects (defined as events requiring medical attention), to be considered safe we expect 0 events of this nature to occur. Additionally, changes in safety questionnaire scores tracking transient within-session changes were considered. Safety questionnaires ask participants to rate commonly experienced symptoms from 0-100 (0= "Not occurring", 100 = "Most severe"). The symptoms assessed are itchiness, tingling, burning sensations, headache, fatigue, nausea, and mood difficulties.
Craniocervical Flexion Test (CCFT) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Fine motor control of neck muscles will be measured via the Craniocervical Flexion Test (CCFT).

SECONDARY OUTCOMES:
European Quality of Life Five Dimension (EQ-5D) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Quality of life will be measured via the European Quality of Life Five Dimension (EQ-5D). Ranges from 0-25 with higher scores indicating reduced quality of life.
Headache Impact Test 6 (HIT-6) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Headache intensity will be measured via the Headache Intensity Test - 6 (HIT-6). This test ranges between a score of 36 and 78 with higher scores meaning increased headache intensity and frequency.
Headache Disability Index (HDI) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Headache effects on participant function will be measured via the Headache Disability Index (HDI). Scores on this index range from 0-100 with higher scores indicating more severe disability as a result of headaches.
Pain Catastrophizing Scale (PCS) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Pain sensitivity will be measured via the Pain Catastrophizing Scale (PCS). Scores on this scale range from 0-52 with higher scores indicating greater sensitivity to pain.
PROMIS Pain Interference Scale | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Patient Reported Outcomes Measurement Information System (PROMIS) Pain interference scale. Ranges from 4-20 with increasing scores meaning increased pain interference in daily life.
Cervical Extensor Endurance Test (CEET) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Neck muscle endurance will be measured via the Cervical Extensor Endurance Test (CEET).
Dynamometry Neck-Strength Assessment (DNSA) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Neck muscle strength will be measured via the Dynamometry Neck-Strength Assessment (DNSA).
Patient health questionnaire 9 (PHQ-9) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Depression will be measured via the patient health questionnaire-9 (PHQ-9). Ranges from 0-27 with higher scores meaning more depressive symptoms.
Generalized anxiety disorder scale 7 (GADS-7) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Anxiety will be measured via the generalized anxiety disorder scale-7 (GADS-7). Ranges from 0-21 with her scores meaning more symptoms of anxiety.
Cervical Flexor Endurance Test (CFET) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Neck muscle endurance will be measured via the Cervical Flexor Endurance Test (CFET) as well.
Numeric Pain Rating Scale (NPRS) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Pain intensity will be assessed through the numeric pain rating scale (NPRS). This scale ranges from 0-10 with a higher score indicating more pain intensity.
Range of Motion of Cervical Joints (ROM) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Range of motion will be assessed through the range of cervical motion test (ROM). A cervical range of motion instrument which measures the angle of cervical motion in each direction (flexion, extension, right and left side bend, right and left rotation over the shoulder) will be used to calculate the total range of motion. This assessment will be pain limited.
Manual Examination of Cervical Joints (MECJ) | To be assessed at baseline, immediately after treatment and at 6 and 12 weeks post treatment.
  Pain at each of the first 3 cervical joints will be assessed through a manual examination of the cervical joints (MECJ). Slight pressure will be applied at each of the first 3 cervical joints (C1/2, C2/3, C3/4) on each side (left and right) by a licensed physiotherapist and participants will be asked to rate their pain from 0-10 at each of these points when pressure is applied with 0 being no pain (more favorable outcome) and 10 being worst possible pain (less favorable outcome).

OTHER OUTCOMES:
Headache Diary | To be completed 2 weeks prior to treatment, 2 weeks after treatment, 2 weeks prior to 6 week assessment, and 2 weeks prior to 12 week assessment for a total of 8 weeks.
  Daily diary for participants to report the frequency, duration, intensity, and location of headaches.
Exercise diary | To be completed each day for the duration of treatment (6 weeks).
  Daily diary for participants to report the intensity and duration of their exercise activities.

CONTACTS AND LOCATIONS:
Overall Officials: Chantel T Debert, MD MSc FRCPC CSCN, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langer L, Levy C, Bayley M. Increasing Incidence of Concussion: True Epidemic or Better Recognition? J Head Trauma Rehabil. 2020 Jan/Feb;35(1):E60-E66. doi: 10.1097/HTR.0000000000000503. PMID 31246881
- [Background] Barnsley L, Lord S, Bogduk N. Whiplash injury. Pain. 1994 Sep;58(3):283-307. doi: 10.1016/0304-3959(94)90123-6. No abstract available. PMID 7838578
- [Background] Sjaastad O, Fredriksen TA, Batnes J, Petersen HC, Bakketeig LS. Whiplash in individuals with known pre-accident, clinical neck status. J Headache Pain. 2006 Feb;7(1):9-20. doi: 10.1007/s10194-006-0270-x. Epub 2006 Feb 20. PMID 16485074
- [Background] Lord SM, Barnsley L, Wallis BJ, Bogduk N. Third occipital nerve headache: a prevalence study. J Neurol Neurosurg Psychiatry. 1994 Oct;57(10):1187-90. doi: 10.1136/jnnp.57.10.1187. PMID 7931379
- [Background] Lindblom U, Verrillo RT. Sensory functions in chronic neuralgia. J Neurol Neurosurg Psychiatry. 1979 May;42(5):422-35. doi: 10.1136/jnnp.42.5.422. PMID 448382
- [Background] Becser N, Sand T, Pareja JA, Zwart JA. Thermal sensitivity in unilateral headaches. Cephalalgia. 1998 Dec;18(10):675-83; discussion 657. doi: 10.1046/j.1468-2982.1998.1810675.x. PMID 9950624
- [Background] Bogduk N, Govind J. Cervicogenic headache: an assessment of the evidence on clinical diagnosis, invasive tests, and treatment. Lancet Neurol. 2009 Oct;8(10):959-68. doi: 10.1016/S1474-4422(09)70209-1. PMID 19747657
- [Background] Bogduk N. Cervicogenic headache: anatomic basis and pathophysiologic mechanisms. Curr Pain Headache Rep. 2001 Aug;5(4):382-6. doi: 10.1007/s11916-001-0029-7. PMID 11403743
- [Background] Dumas JP, Arsenault AB, Boudreau G, Magnoux E, Lepage Y, Bellavance A, Loisel P. Physical impairments in cervicogenic headache: traumatic vs. nontraumatic onset. Cephalalgia. 2001 Nov;21(9):884-93. doi: 10.1046/j.1468-2982.2001.00264.x. PMID 11903282
- [Background] Manchikanti L, Pampati V, Kaye AD, Hirsch JA. Cost Utility Analysis of Cervical Therapeutic Medial Branch Blocks in Managing Chronic Neck Pain. Int J Med Sci. 2017 Oct 15;14(13):1307-1316. doi: 10.7150/ijms.20755. eCollection 2017. PMID 29200944
- [Background] Frazer A, Williams J, Spittles M, Rantalainen T, Kidgell D. Anodal transcranial direct current stimulation of the motor cortex increases cortical voluntary activation and neural plasticity. Muscle Nerve. 2016 Nov;54(5):903-913. doi: 10.1002/mus.25143. Epub 2016 May 20. PMID 27065472
- [Background] Rroji O, van Kuyck K, Nuttin B, Wenderoth N. Anodal tDCS over the Primary Motor Cortex Facilitates Long-Term Memory Formation Reflecting Use-Dependent Plasticity. PLoS One. 2015 May 21;10(5):e0127270. doi: 10.1371/journal.pone.0127270. eCollection 2015. PMID 25996937
- [Background] Zaninotto AL, El-Hagrassy MM, Green JR, Babo M, Paglioni VM, Benute GG, Paiva WS. Transcranial direct current stimulation (tDCS) effects on traumatic brain injury (TBI) recovery: A systematic review. Dement Neuropsychol. 2019 Apr-Jun;13(2):172-179. doi: 10.1590/1980-57642018dn13-020005. PMID 31285791
- [Background] Wessel MJ, Zimerman M, Hummel FC. Non-invasive brain stimulation: an interventional tool for enhancing behavioral training after stroke. Front Hum Neurosci. 2015 May 15;9:265. doi: 10.3389/fnhum.2015.00265. eCollection 2015. PMID 26029083
- [Background] O'Connell NE, Marston L, Spencer S, DeSouza LH, Wand BM. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2018 Apr 13;4(4):CD008208. doi: 10.1002/14651858.CD008208.pub5. PMID 29652088
- [Background] Begemann MJ, Brand BA, Curcic-Blake B, Aleman A, Sommer IE. Efficacy of non-invasive brain stimulation on cognitive functioning in brain disorders: a meta-analysis. Psychol Med. 2020 Nov;50(15):2465-2486. doi: 10.1017/S0033291720003670. Epub 2020 Oct 19. PMID 33070785
- [Background] Stilling JM, Monchi O, Amoozegar F, Debert CT. Transcranial Magnetic and Direct Current Stimulation (TMS/tDCS) for the Treatment of Headache: A Systematic Review. Headache. 2019 Mar;59(3):339-357. doi: 10.1111/head.13479. Epub 2019 Jan 23. PMID 30671941
- [Background] Rahimi MD, Fadardi JS, Saeidi M, Bigdeli I, Kashiri R. Effectiveness of cathodal tDCS of the primary motor or sensory cortex in migraine: A randomized controlled trial. Brain Stimul. 2020 May-Jun;13(3):675-682. doi: 10.1016/j.brs.2020.02.012. Epub 2020 Feb 14. PMID 32289696
- [Background] Andrade SM, de Brito Aranha REL, de Oliveira EA, de Mendonca CTPL, Martins WKN, Alves NT, Fernandez-Calvo B. Transcranial direct current stimulation over the primary motor vs prefrontal cortex in refractory chronic migraine: A pilot randomized controlled trial. J Neurol Sci. 2017 Jul 15;378:225-232. doi: 10.1016/j.jns.2017.05.007. Epub 2017 May 3. PMID 28566169
- [Background] Dunning JR, Butts R, Mourad F, Young I, Fernandez-de-Las Penas C, Hagins M, Stanislawski T, Donley J, Buck D, Hooks TR, Cleland JA. Upper cervical and upper thoracic manipulation versus mobilization and exercise in patients with cervicogenic headache: a multi-center randomized clinical trial. BMC Musculoskelet Disord. 2016 Feb 6;17:64. doi: 10.1186/s12891-016-0912-3. PMID 26852024
- [Background] Fernandez M, Moore C, Tan J, Lian D, Nguyen J, Bacon A, Christie B, Shen I, Waldie T, Simonet D, Bussieres A. Spinal manipulation for the management of cervicogenic headache: A systematic review and meta-analysis. Eur J Pain. 2020 Oct;24(9):1687-1702. doi: 10.1002/ejp.1632. Epub 2020 Jul 20. PMID 32621321
- [Background] Chaibi A, Russell MB. Manual therapies for cervicogenic headache: a systematic review. J Headache Pain. 2012 Jul;13(5):351-9. doi: 10.1007/s10194-012-0436-7. Epub 2012 Mar 30. PMID 22460941
- [Background] Debarnot U, Neveu R, Samaha Y, Saruco E, Macintyre T, Guillot A. Acquisition and consolidation of implicit motor learning with physical and mental practice across multiple days of anodal tDCS. Neurobiol Learn Mem. 2019 Oct;164:107062. doi: 10.1016/j.nlm.2019.107062. Epub 2019 Aug 1. PMID 31377178
- [Background] Lefebvre S, Laloux P, Peeters A, Desfontaines P, Jamart J, Vandermeeren Y. Dual-tDCS Enhances Online Motor Skill Learning and Long-Term Retention in Chronic Stroke Patients. Front Hum Neurosci. 2013 Jan 9;6:343. doi: 10.3389/fnhum.2012.00343. eCollection 2012. PMID 23316151
- [Background] Hatem SM, Saussez G, Della Faille M, Prist V, Zhang X, Dispa D, Bleyenheuft Y. Rehabilitation of Motor Function after Stroke: A Multiple Systematic Review Focused on Techniques to Stimulate Upper Extremity Recovery. Front Hum Neurosci. 2016 Sep 13;10:442. doi: 10.3389/fnhum.2016.00442. eCollection 2016. PMID 27679565
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Cote P, Yu H, Shearer HM, Randhawa K, Wong JJ, Mior S, Ameis A, Carroll LJ, Nordin M, Varatharajan S, Sutton D, Southerst D, Jacobs C, Stupar M, Taylor-Vaisey A, Gross DP, Brison RJ, Paulden M, Ammendolia C, Cassidy JD, Loisel P, Marshall S, Bohay RN, Stapleton J, Lacerte M. Non-pharmacological management of persistent headaches associated with neck pain: A clinical practice guideline from the Ontario protocol for traffic injury management (OPTIMa) collaboration. Eur J Pain. 2019 Jul;23(6):1051-1070. doi: 10.1002/ejp.1374. Epub 2019 Feb 28. PMID 30707486
- [Background] Rani M, Kaur J. Effectiveness of different physiotherapy interventions in the management of cervicogenic headache: a pilot randomized controlled trial. J Man Manip Ther. 2022 Apr;30(2):96-104. doi: 10.1080/10669817.2021.1962687. Epub 2021 Aug 10. PMID 34374330
- [Background] Houts CR, McGinley JS, Wirth RJ, Cady R, Lipton RB. Reliability and validity of the 6-item Headache Impact Test in chronic migraine from the PROMISE-2 study. Qual Life Res. 2021 Mar;30(3):931-943. doi: 10.1007/s11136-020-02668-2. Epub 2020 Oct 20. PMID 33079313
- [Background] Eyres S, Carey A, Gilworth G, Neumann V, Tennant A. Construct validity and reliability of the Rivermead Post-Concussion Symptoms Questionnaire. Clin Rehabil. 2005 Dec;19(8):878-87. doi: 10.1191/0269215505cr905oa. PMID 16323387
- [Background] Jabbari S, Salahzadeh Z, Sarbakhsh P, Rezaei M, Farhoudi M, Ghodrati M. Validity and Reliability of Persian Version of Henry Ford Hospital Headache Disability Inventory Questionnaire. Arch Iran Med. 2021 Oct 1;24(10):752-758. doi: 10.34172/aim.2021.111. PMID 34816697
- [Background] Robinson-Papp J, George MC, Wongmek A, Nmashie A, Merlin JS, Ali Y, Epstein L, Green M, Serban S, Sheth P, Simpson DM. The Quantitative Analgesic Questionnaire: A Tool to Capture Patient-Reported Chronic Pain Medication Use. J Pain Symptom Manage. 2015 Sep;50(3):381-6. doi: 10.1016/j.jpainsymman.2015.03.013. Epub 2015 Apr 23. PMID 25912277
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244
- [Background] James G, Doe T. The craniocervical flexion test: intra-tester reliability in asymptomatic subjects. Physiother Res Int. 2010 Sep;15(3):144-9. doi: 10.1002/pri.456. PMID 20146239
- [Background] Sebastian D, Chovvath R, Malladi R. Cervical extensor endurance test: a reliability study. J Bodyw Mov Ther. 2015 Apr;19(2):213-6. doi: 10.1016/j.jbmt.2014.04.014. Epub 2014 Apr 18. PMID 25892374
- [Background] Versteegh T, Beaudet D, Greenbaum M, Hellyer L, Tritton A, Walton D. Evaluating the reliability of a novel neck-strength assessment protocol for healthy adults using self-generated resistance with a hand-held dynamometer. Physiother Can. 2015 Winter;67(1):58-64. doi: 10.3138/ptc.2013-66. PMID 25931654
- [Background] Cleland BT, Galick M, Huckstep A, Lenhart L, Madhavan S. Feasibility and Safety of Transcranial Direct Current Stimulation in an Outpatient Rehabilitation Setting After Stroke. Brain Sci. 2020 Oct 9;10(10):719. doi: 10.3390/brainsci10100719. PMID 33050340
- [Background] Osman A, Barrios FX, Kopper BA, Hauptmann W, Jones J, O'Neill E. Factor structure, reliability, and validity of the Pain Catastrophizing Scale. J Behav Med. 1997 Dec;20(6):589-605. doi: 10.1023/a:1025570508954. PMID 9429990
- [Background] Stark RG, Reitmeir P, Leidl R, Konig HH. Validity, reliability, and responsiveness of the EQ-5D in inflammatory bowel disease in Germany. Inflamm Bowel Dis. 2010 Jan;16(1):42-51. doi: 10.1002/ibd.20989. PMID 19475674
- [Background] Harris KD, Heer DM, Roy TC, Santos DM, Whitman JM, Wainner RS. Reliability of a measurement of neck flexor muscle endurance. Phys Ther. 2005 Dec;85(12):1349-55. PMID 16305273
- [Derived] Jobin K, Campbell C, Schabrun SM, Schneider KJ, Smith A, Debert CT. The safety and feasibility of transcranial direct current stimulation combined with conservative treatment for patients with cervicogenic headaches: A double-blinded randomized control study protocol. Contemp Clin Trials Commun. 2024 Sep 19;42:101370. doi: 10.1016/j.conctc.2024.101370. eCollection 2024 Dec. PMID 39391228